CLINICAL TRIAL: NCT03168685
Title: Bayer/HITLAB - Hemophilia Mobile App Usability Pilot
Brief Title: Hemophilia Mobile App Usability Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Healthcare Innovation Technology Lab (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00021564
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hemophilia
Keywords: smartphones; clinical trials; weight; actigraph; tracking; hemophilia
MeSH Terms: conditions — Hemophilia A; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental (Experimental): Multiple device intervention
  1. SureSource Engage mobile application
  2. ActiGraph Link
  3. weight scale
  Interventions: Device: SureSource Engage application

INTERVENTIONS:
Device: SureSource Engage application — Eligible patients who choose to participate in the study will be asked to wear an actigraphy device [ActiGraph GT9X Link "Actigraph Link"] on their wrist continuously during both 4-week study phases.
  The ActiGraph Link is a small (3.5 X 3.5 X 1 cm) wristwatch like device weighing approximately 14 grams that measures indicators of the wearer's activity and sleep patterns, including: acceleration, energy expenditure, steps, basal metabolic rate, activity intensity, sleep time, sleep efficiency, sleep latency, and body position.
  The application being utilized is SureSource Engage application from Clinical Ink. The application is compatible to most Android and iOS devices.
  Participants will also use a basic Bluetooth-enabled weight scale that syncs with the application.
  Other Names: ActiGraph GT9X Link; weight scale

SUMMARY:
The purpose of this study is to evaluate the utility and user experience of a smart phone app for people with medical conditions, used in conjunction with an ActiGraph wearable device and a connected scale.

DETAILED DESCRIPTION:
HITLAB will conduct a segmented rapid user acceptance study ("rapid UX study") of a smart phone app and an actigraphy device with a connected scale. During the first segment, of one month's duration, subjects will use the app, actigraphy device, and scale. Next, over an interphase period of up to 6 weeks, subjects will only use the app. During this time, the app will be modified based on data collected during the first segment. Finally, during the second period, also of one month's duration, subjects will use the modified app, actigraphy device, and scale.

ELIGIBILITY:
Inclusion Criteria:

1. You own an iPhone or a Samsung (S5 or higher) smartphone
2. Your age is between 18 and 63 years
3. You reside in the New York metropolitan area
4. You are able to read, write, and speak English
5. You have participated in a concluded clinical trial in the past two years

Exclusion Criteria:

1. You do not own an iPhone or a Samsung (S5 or higher) smartphone
2. Your age is not between 18 and 63 years
3. You do not reside in the New York metropolitan area
4. You are not able to read, write, and speak English
5. You have not participated in a concluded clinical trial in the past two years

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-05-11 (Estimated); Study Completion 2018-05-11 (Estimated)

PRIMARY OUTCOMES:
Usage of the SureSource Engage application as assessed by ActiLife software | 128 days
Device usability as assessed by the System Usability Scale (SUS) | 128 days

CONTACTS AND LOCATIONS:
Overall Officials: Stan Kachnowski, PhD, MPA, Principal Investigator — Healthcare Innovation Technology Lab; Ryan Dammerman, MD, Principal Investigator — Healthcare Innovation Technology Lab
Locations (1):
- Healthcare Innovation and Technology Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No